## Date:26/11/2016

## Informed Consent

I agree to participate in this study titled:

Comparison of Recurrence Rate of Ferguson Gross Herniotomy with Mitchell Banks
Herniotomy in Children Older than 2 years.

The doctor has told me that my child is suffering from hernia which can be operated by Mitchell Banks Technique or Fergusson Gross Technique. The merits and demerits of both these techniques have been well explained to me and I have read them as well which were provided to me in separate brochure.

I understand that I am free to withdraw from the study whenever I want to and I have been told by doctors that they will continue to give my child the best possible care even after my discontinuation of study.

Furthermore, I allow the researcher or any other person authorized by the researcher to contact me at my home or an address given by me for the treatment and follow up. I have been assured that the information provided by me will be kept confidential and will be used for research purpose only.

| Patient Name: | Witness Name: |
|-------------------------|---------------|
| CNIC No: | CNIC No: |
| Signature: | Signature: |
| Date: | Date: |
| Investigator signature: | |
| Date: | |